CLINICAL TRIAL: NCT01376180
Title: Drug Use Investigation for LAMICTAL
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112727
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed lamotrigine tablet: Subjects with epilepsy prescribed lamotrigine tablet during study period
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Administered according to the prescribing information in the locally approved label by the authorities

SUMMARY:
The purpose of this study is to grasp actual status of usage of lamotrigine tablet and to collect information for using lamotrigine tablet effectively and safely as well as to grasp onset status of adverse events in pediatric subjects, geriatric subjects, pregnant women, subjects with poor renal and hepatic functions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with epilepsy having the following seizure types.
* Partial seizures (including secondary generalized seizures)
* Tonic-clonic seizures
* Generalized seizures of Lennox-Gastaut syndrome

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with epilepsy having the following seizure types.
  * partial seizures (including secondary generalized seizures)
  * tonic-clonic seizures
  * generalized seizures of Lennox-Gastaut syndrome
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2008-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects with epilepsy treated with lamotrigine tablet | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Sunao Kaneko, Yushi Inoue, Masafumi Iijima, Atsuko Ishida, Shogo Inoshiri. Drug Use Investigation of Lamotrigine Tablets in Patients with Epilepsy - Results of Interim Analysis -. 2011;60(3):9-35.